CLINICAL TRIAL: NCT01918098
Title: A Randomized, Double-blind, Double-dummy, Parallel-group, Multicenter Study to Demonstrate Improvement in Symptoms of Constipation in Subjects With Moderate to Severe Non-malignant Pain Taking Oxycodone Equivalent of ≥10 mg/Day and ≤50 mg/Day as Oxycodone/Naloxone Prolonged-release (OXN) Compared to Subjects Taking Oxycodone Prolonged-release (OXY) Tablets Alone.
Brief Title: Targin for Non-cancer Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma (China) Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OXN08-CN-302a
Record Dates: First submitted 2013-08-05; First posted 2013-08-07 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Non Cancer Pain
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxycodone/naloxone prolonged release tablets (Experimental): Dose strength:5/2.5 mg,10/5mg, 20/10mg,PO,q12h.daily dose from 10/5mg to 50/25mg.treatment duration:12 weeks
  Interventions: Drug: Oxycodone/naloxone prolonged release tablets
- Oxycodone prolonged release tablets (Active Comparator): Dose strength:5mg,10mg, 20mg,PO,q12h.daily dose from 10mg to 50mg.treatment duration:12 weeks
  Interventions: Drug: Oxycodone/naloxone prolonged release tablets

INTERVENTIONS:
Drug: Oxycodone/naloxone prolonged release tablets

SUMMARY:
To determine the improvement in symptoms of constipation in subjects receiving treatment with oxycodone/naloxone prolonged release tablets (OXN) compared to oxycodone prolonged release tablets (OXY) based on the Bowel Function Index (BFI)

ELIGIBILITY:
Screening Inclusion criteria:

* Males or females, 18 years of age or older
* Clinical diagnosis of musculo-skeletal pain for 4 weeks or longer with non-malignant pain etiology at Visit 1. Possible etiologies are conditions related to intervertebral disc disease, spondylolisthesis and osteoarthritis; other similar non-malignant diseases are also eligible.
* Patients with non-malignant pain that require around-the-clock opioid therapy (oxycodone equivalent of ≥10 mg/day and ≤50 mg/day) who are likely to benefit from WHO step III opioid therapy for the duration of the study
* Patients who have been already treated with NSAIDs at least 2 weeks before enrolment are also eligible, but they should rate their pain (Pain Intensity Scale -"average pain" over the last 24 hours) as ≥4 on 0-10 scale."
* Subjects are either taking opioid medication or willing to take opioids to treat their pain
* Patients who are willing to use adequate and reliable contraception throughout the study. Highly effective methods of birth control are defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as sterilization, implants, injectable, combined oral contraceptives, some IUDs (intrauterine Device, hormonal), sexual abstinence or vasectomized partner
* Subjects willing and able to participate in all aspects of the study, including use of oral medication, completion of subjective evaluations, attending scheduled clinic visits, completing telephone contacts, and compliance with protocol requirements are evidenced by providing written informed consent
* Subjects taking pre-study, non-opioid analgesics, and all other concomitant medications, including those medications for the treatment of depression and are considered necessary for the subject's welfare, and are anticipated to remain stable throughout the double-blind period of the study, and are to be continued under the supervision of the investigator, are eligible.

  * Patients who have been already treated with NSAIDs at least 2 weeks before enrolment are also eligible, but they should rate their pain (Pain Intensity Scale -"average pain" over the last 24 hours) as ≥4 on 0-10 scale.

Criteria for entry to the Double-Blind phase:

1. Subjects continue to satisfy screening criteria outlined in the protocol
2. Subject's OXY dose is between 10-50 mg/day
3. Subjects who rate their pain (Pain Intensity Scale -"average pain" over the last 24 hours) as≤4 on 0-10 scale with less than or equal to two doses of Morphine Sulfate tablets rescue medication per day for either the last three consecutive days or four of the last seven days
4. Subjects who have constipation induced, or worsened by their opioid study medication, as shown by:

   1. The subject's medical need for regular intake of laxatives to have at least 3 bowel evacuations per week, or having less than 3 bowel evacuations per week when not taking a laxative, respectively and
   2. The subjects' constipation was considered to be induced, worsened or maintained by their current study opioid medication and
   3. BFI value > 30.
5. Subjects demonstrate compliance with laxative use, and completing appropriate and legible daily diaries
6. Subjects taking daily fibre supplementation or bulking agents are eligible if they can be maintained on a stable dose and regimen throughout the study, and in the investigator's opinion are willing and able to maintain adequate hydration.

Screening Exclusion criteria:

1. Females who are pregnant (positive β-hCG test) or lactating
2. Any history of hypersensitivity or with any contraindication to oxycodone, naloxone, bisacodyl, or related products
3. Subjects currently taking the equivalent of > 50 mg/day Oxycodone PR
4. Evidence of clinically significant cardiovascular, renal, hepatic, gastrointestinal (paralytic ileus), or psychiatric disease, as determined by medical history, clinical laboratory tests, electrocardiogram (ECG) results, and physical examination, that will place the subject at risk upon exposure to the study medication or that could confound the analysis and/or interpretation of the study results
5. Subjects with evidence of impaired liver/kidney function upon entry into the study defined as aspartate aminotransferase (AST; SGOT), alanine aminotransferase (ALT; SGPT), or alkaline phosphatase levels >3 times the upper limit of normal; gamma glutamyltranspeptidase (GGT or GGTP) ≥ 5 times the upper limit of normal; total bilirubin level outside of the reference range; and/or creatinine level outside of the reference range or >2 mg/dl, or in the investigator's opinion, liver and/or kidney impairment to the extent that the subject should not participate in this study
6. Subjects with evidence of significant structural abnormalities of the gastrointestinal tract or any diseases/conditions that affect bowel transit
7. Subjects who have required treatment for the diagnosis of irritable bowel syndrome (IBS)
8. Subjects receiving hypnotics or other central nervous system (CNS) depressants that, in the investigator's opinion, may pose a risk of additional CNS depression with opioids study medication
9. Surgery within 2 months prior to the start of the Screening Period, or planned surgery during the 12-week Double-blind Phase that may have affected GI motility or pain
10. Subjects diagnosed with cancer, not including basal cell carcinoma
11. Subjects with Rheumatoid Arthritis (RA)
12. Subjects receiving opioid substitution therapy for opioid addiction (e.g., methadone or buprenorphine)
13. Subjects with active alcohol or drug abuse and/or history of opioid abuse
14. Subjects who participated in a clinical research study involving a new chemical entity or an experimental drug within 30 days of study entry (defined as the start of the Screening Period)
15. Subjects presently taking, or who had taken naloxone or naltrexone within 30 days of study entry (defined as the start of the Screening Period).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Bowel function index(BFI) 12 Weeks | 12 weeks

SECONDARY OUTCOMES:
Modified BPI-SF-Average Pain over the last 24 hours | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Yu, Study Director — Mundipharma, China
Locations (31):
- China (31):
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Second Affiliated Hospital of Shan Tou University Medical College, Shantou, Guangdong
  - Hebei General Hospital, Shijiazhuang, Hebei
  - Beijing friendship hospital, Beijing
  - Beijing Tiantan Hospital, Beijing
  - Beijing Union hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The first affiliated hospital of Bengbu medical collage, Bengbu
  - The third Xiangya hospital of central south university, Changsha
  - The thrid Xiangya Hospital of central south university, Changsha
  - Xiangya hospital central south university, Changsha
  - West China Hospital, Chengdu
  - Daping Hospital, Chongqing
  - South West hospital, Chongqing
  - Fuzhou general hospital, Fuzhou
  - The third affiliated hospital Sun yat-sen university, Guangzhou
  - Guizhou Provincial People's Hospital, Guizhou
  - The second affiliated hospital of Harbin medical university, Harbin
  - Shandong Provincial Hospital, Jinan
  - Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai Changhai Hospital, Shanghai
  - Shanghai Sixth People's Hospital, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - The first affiliated hospital of Shantou university medical college, Shantou
  - The general hospital of Shenyang military, Shenyang
  - The central hospital of Wuhan, Wuhan
  - Tongji Hospital, Wuhan
  - Union Hospital Tongji medical college, Wuhan
  - The affiliated hospital of Xuzhou medical university, Xuzhou
  - Second affiliated hospital of Zhejiang university, Zhejiang

REFERENCES:
- [Derived] Leng X, Zhang F, Yao S, Weng X, Lu K, Chen G, Huang M, Huang Y, Zeng X, Hopp M, Lu G. Prolonged-Release (PR) Oxycodone/Naloxone Improves Bowel Function Compared with Oxycodone PR and Provides Effective Analgesia in Chinese Patients with Non-malignant Pain: A Randomized, Double-Blind Trial. Adv Ther. 2020 Mar;37(3):1188-1202. doi: 10.1007/s12325-020-01244-x. Epub 2020 Feb 3. PMID 32020565